CLINICAL TRIAL: NCT03609489
Title: Apatinib Combined Capecitabine Versus Capecitabine Alone for Adjuvant Therapy in Patients After Biliary Carcinoma Surgery: a Prospective Randomized Controlled Study
Brief Title: A Study to Investigate Apatinib Combined Capecitabine on Adjuvant Therapy of Biliary Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jie Ma, Deputy director, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRGX05
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Biliary Carcinoma
Keywords: Biliary cancer; adjuvant therapy; apatinib; capecitabine
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Apatinib combined with Capetabine
  Interventions: Drug: Capecitabine; Drug: Apatinib
- Control Group (Active Comparator): Capecitabine
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine, 1000mg/m2, oral administration, twice daily (once in the morning and once in the evening with an interval of 12 hours, equivalent to a total daily dose of 2000 mg/m2), continuous medication for 14 days and off for 7 days. Every 21 days is a cycle, and there shall be a total of 8 cycles. If the subject is still unable to tolerate toxicity after experiencing two dose adjustments, he/she should be moved out of the group.
  Other Names: Xeloda
Drug: Apatinib — Apatinib, 500 mg, administered orally (after breakfast) once daily from day 1 to day 21 (including day 21) with continuous administration. Every 21 days serve as a cycle. If after 2 dose adjustments, the subject is still unable to tolerate toxicity, he/she should be moved out of the group.
  Other Names: Aitan
  Arms: Test Group

SUMMARY:
It is a prospective,parallel study to investigate the saftety and efficacy of Apatinib combined Capacitabine in the adjuvant treatment of the biliary cancinoma after operation.

DETAILED DESCRIPTION:
Subjects were randomly divided into experimental and control groups. The experimental group was postoperatively treated with apatinib combined with capecitabine for adjuvant therapy of biliary cancer, and the control group was treated with capecitabine alone.

Progression free survival (PFS), overall survival (OS), time to progression (TTP), objective response rate (ORR), disease control rate (DCR), EORTC QLQ-C30, HCC-18 and drug safety: vital signs, laboratory indicators, adverse event (AE), and serious adverse event (SAE), drug-related AE and SAE and their specific AE (such as hypertension, proteinuria, and hand-foot syndrome) were followed for research in the two groups to evaluate the efficacy and safety of the two regimens for the treatment of biliary tract cancer according to the standard of NCI-CTCAE V4.0.

A rigorous, randomized and prospective study was conducted to compare the efficacy and safety in treating biliary cancer between the combined use of apatinib mesylate plus capecitabine and capecitabine alone, with a view to improving the survival outcome and life quality of patients with biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fully aware of the research and voluntarily signed informed consent (informed consent must be signed prior to the execution of any required test procedure);
* Patients received removal of biliary tract cancers that have been confirmed by histology or cytology, including intrahepatic bile duct carcinoma (IHCC), extrahepatic bile duct cancer (EHCC), and gallbladder cancer(GBC);
* Normal function of major organs that meets the following criteria:

Blood routine examination:

HB≥90 g/L； ANC≥1.5×109/L； PLT≥60×109/L；

Biochemical examination:

ALB ≥29 g/L； ALT and AST<2.5ULN； TBIL ≤2ULN； Creatinine≤1.5ULN;

* ECOG physical condition scores 0 or 1;
* Fertile male or female patients volunteer to use effective contraception methods during the research period, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc.
* Fertile and non-lactational female who show negative in serum or urine pregnancy test within 7 days before inclusion for the study.

Exclusion Criteria:

* Those who received approved or on-going anti-tumor therapy within 4 weeks before the research;
* Those who received other anti-angiogenic tyrosine kinase inhibitors or monoclonal antibodies that had been approved or under study before the research;
* Abnormal laboratory tests that have significant clinical implication;
* International normalized ratio (INR) ≥ 1.5 or partially activated prothrombin time (APTT) ≥ 1.5 × ULN;
* The patient's current serum potassium, serum magnesium, or serum calcium is below the normal reference range of laboratory test (whether supplemented or not), or >CTCAE grade 1;
* Patients currently suffering from hypertension that cannot be controlled with drugs;
* The researchers conclude electrolyte abnormalities that are clinically significant;
* There is severe bleeding or hemoptysis in the past or at current stage, or there are thromboembolic events within 12 months;
* Cardiovascular diseases that are clinically significant;
* ECG showed QTcB interval ≥ 480 milliseconds in resting state;
* Suffering from other malignant tumors in the past 5 years, excluding basal cell carcinoma or squamous cell carcinoma after receiving radical surgery, or carcinoma in situ of cervix;
* Active or uncontrollable serious infection (≥ CTCAE grade 2 infection), including but not limited to human immunodeficiency virus (HIV) infection;
* Known history of liver disease with evident significance;
* The patient currently has brain metastasis or spinal compression, except individual cases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  the length of time during the recruiment and after the progression of the biliary cancer verified by imagine examination

SECONDARY OUTCOMES:
overall survival | 24 months
  the length of time during the recruitment and after the death of the patient
objective response rate | 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response and partial response cases
Disease Control rate | 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response, partial response and stable disease cases

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ma, doctor, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Luvira V, Satitkarnmanee E, Pugkhem A, Kietpeerakool C, Lumbiganon P, Pattanittum P. Postoperative adjuvant chemotherapy for resectable cholangiocarcinoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD012814. doi: 10.1002/14651858.CD012814.pub2. PMID 34515993